CLINICAL TRIAL: NCT00451854
Title: Student Athlete Drug Surveillance Trail
Brief Title: Student Athlete Testing Using Random Notification
Acronym: SATURN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA-12018
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2007-03

CONDITIONS: Drug Abuse; Alcohol Abuse; Substance Abuse
Keywords: Drug testing; Adolescence; Student athlete; Substance abuse; Alcohol use; Drug use
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Alcohol Drinking | interventions — Random Allocation; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Random, no advanced notice drug and alcohol testing

SUMMARY:
The purpose of this study is to determine the influence of drug testing on risk and protective factors of substance abuse among adolescents; examine whether drug and alcohol testing among high school athletes leads to reduced drug and alcohol use; and assess the use of drugs and alcohol among student athletes and non-athletes.

DETAILED DESCRIPTION:
This proposal is designed to address the increase in drug use among adolescent athletes by studying a school-based version of the random, no-advance warning drug testing program used by the United States Olympic Committee (USOC). High school athletes are a large group, comprising 50% of their school's enrollment. They have a high rate of substance abuse behaviors similar to the general school population, and an even higher use of 'ergrogenic' (athletic enhancing) drugs. Recognizing the high rate of substance abuse among young athletes and their 'role model' effect on other students, the U.S. Supreme Court recently upheld an Oregon School Districts' policy to randomly drug test students engaged in school-sponsored sports. Drug testing has the potential to deter adolescent substance abuse. It is gender-neutral, without ethnic bias and provides a potentially powerful environmental influence. However, despite its legality and theorized effectiveness, schools are implementing drug surveillance without the benefit of randomized, prospective efficacy research.

Focusing on adolescent athletes provides a unique opportunity to study the prevention effect of drug testing. All sports teams in 24 schools who agree to implement mandatory testing as school policy but have never implemented this policy, will be randomly assigned by school, to three years of either: 1) random, no-advance warning drug testing or 2) a 3-year control period without testing. Selection of students for drug testing will be random, with no exclusions for having been previously tested. State-of-the-art testing will include physician specimen collectors under the direction of research physicians (PI & Co-I), who are Certified USOC Drug Surveillance Crew Chiefs, with specimen analysis at the UCLA Olympic Laboratory using the most accurate analytical techniques to minimize false negative (reducing policy integrity) and false positive (mislabeling students) results. Confidential questionnaires will be completed by student-athletes twice yearly to assess risk and protective factors for drug use and assess self-reported substance abuse. The role model effect of the surveillance program on nonathletes' drug use will be assessed twice yearly by anonymous survey. We will determine the effect of drug testing policy on: 1) adolescent drug use mediators, 2) actual drug use behaviors of student-athletes and their non-athlete peers, and 3) potential gender and demographic differences. Reliability of subjective questionnaire responses will be assessed by comparisons with objective drug test results. Study findings will assist school districts and education agencies evaluate, guide, and implement future drug prevention policy decisions.

ELIGIBILITY:
Inclusion Criteria:

- Schools without previous drug and alcohol testing policies, willing to design and implement a drug and alcohol policy conforming to the United States Supreme Court Decision (Acton v Vernonia, willing to be randomized to an active drug testing or control (deferred testing) condition, and agreement of school district school board and principals

Exclusion Criteria:

- Schools with current alcohol or drug testing policy, unwillingness to be randomized to control and drug testing

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14000
Dates: Start 1999-09; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
The specific measure that will be used to determine the effect of the intervention on drug and alcohol use as determined by confidential and anonymous surveys.

SECONDARY OUTCOMES:
Potential risk and protective factors for drug and alcohol use behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Linn Goldberg, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Divsion of Health Promotion & Sports Medicine, Portland, Oregon, United States

REFERENCES:
- [Result] Goldberg L, Elliot DL, MacKinnon DP, Moe E, Kuehl KS, Nohre L, Lockwood CM. Drug testing athletes to prevent substance abuse: background and pilot study results of the SATURN (Student Athlete Testing Using Random Notification) study. J Adolesc Health. 2003 Jan;32(1):16-25. doi: 10.1016/s1054-139x(02)00444-5. PMID 12507797
- [Derived] Goldberg L, Elliot DL, MacKinnon DP, Moe EL, Kuehl KS, Yoon M, Taylor A, Williams J. Outcomes of a prospective trial of student-athlete drug testing: the Student Athlete Testing Using Random Notification (SATURN) study. J Adolesc Health. 2007 Nov;41(5):421-9. doi: 10.1016/j.jadohealth.2007.08.001. PMID 17950161